CLINICAL TRIAL: NCT06600061
Title: Bilateral Erector Spinae Plane Block as an Opioid Sparing Technique for Selective Dorsal Rhizotomy in Pediatric Patients With Spastic Cerebral Palsy: A Randomized Controlled Trial
Brief Title: Bilateral Erector Spinae Plane Block as an Opioid Sparing Technique for Selective Dorsal Rhizotomy in Pediatric Patients With Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR838/9/24
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Erector Spinae Plane Block; Opioid; Sparing; Selective Dorsal Rhizotomy; Pediatric; Spastic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block group (Experimental): Patients will receive erector spinae plane block after induction of anesthesia.
  Interventions: Other: Erector Spinae Plane Block
- Control group (No Intervention): Patients will not receive erector spinae plane block.

INTERVENTIONS:
Other: Erector Spinae Plane Block — Patients will receive erector spinae plane block after induction of anesthesia.
  Arms: Erector Spinae Plane Block group

SUMMARY:
This study aims to evaluate the efficacy of bilateral erector spinae plane block as an opioid-sparing technique for selective dorsal rhizotomy in pediatric patients with spastic cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common physical disability affecting children. Selective dorsal rhizotomy (SDR) is a neurosurgical procedure that permanently reduces lower limb spasticity in children with CP by selectively targeting and removing sensory rootlets with aberrant activity.

Postoperative pain is often distressing for patients and their families and can result in complications, delayed participation in therapy, and poor functional recovery. Erector spinae plane block (ESPB) is a newly described interfascial plane block. ESPB is effective on both visceral and somatic pain.

ELIGIBILITY:
Inclusion Criteria:

* Age from 6 to 18 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status II, III.
* Patients with spastic cerebral palsy undergoing selective dorsal rhizotomy.

Exclusion Criteria:

* Allergy to local anesthetics.
* Severe fixed joint deformity.
* Previous orthopedic surgery.
* Patient with abnormal liver/kidney function.
* Patient with skin damage or infection at the proposed puncture site.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia of 0.05 mg/kg morphine will be given if the Wong-Baker score is 4 more to be repeated after 30 min if pain persists until the Wong-Baker score < 4.

SECONDARY OUTCOMES:
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from end of surgery to the first dose of morphine administrated) will be assessed.
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the Wong-Baker pain rating scale (The scale contains a series of six faces ranging from a happy face at 0 to indicate "no hurt" to a crying face at 10 to indicate "hurts worst"). Wong-Baker score will be assessed at post anesthesia care unit, 4, 6, 8, 12, 18 and 24 h postoperatively.
Patient satisfaction | 24 hours postoperatively
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied)
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as Local anesthetic systemic toxicity (LAST), bradycardia, hypotension, postoperative nausea and vomiting (PONV), respiratory depression, or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.